CLINICAL TRIAL: NCT02075203
Title: A Randomized, Placebo Controlled, Partially Blinded Phase II Study to Evaluate Safety, Immunogenicity, and Prevention of Infection With Mycobacterium Tuberculosis of AERAS-404 and BCG Revaccination in Healthy Adolescents
Brief Title: Evaluation of Safety, Immunogenicity, and Prevention of TB With AERAS-404 and BCG Revaccination in Healthy Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aeras (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C-040-404
Record Dates: First submitted 2014-02-17; First posted 2014-03-03 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-05

CONDITIONS: Tuberculosis
Keywords: BCG Vaccinated
MeSH Terms: conditions — Tuberculosis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AERAS-404 (15 mcgH4/500 nmol IC31) (Experimental): 2 doses on Study Days 0 and 56
  Interventions: Biological: AERAS-404
- Bacillus Calmette-Guérin (BCG) (Active Comparator): 1 Dose on Study Day 0
  Interventions: Biological: Bacillus Calmette-Guérin (BCG)
- Placebo (Placebo Comparator): 2 Doses on Study Days 0 and 56
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: AERAS-404 — The H4 antigen is a fusion protein created from two Mtb antigens: antigen Ag85B and TB10.4. Ag85B is also referred to as α-antigen and is a 30-kDa mycolyl transferase protein. TB10.4 is one of three members of the very similar ESAT-6 group of proteins found in Mtb culture supernatants. TB10.4 induces broad immune responses in T cells isolated from TB subjects compared to BCG-vaccinated donors and unvaccinated donors. IC31 is a combination of a leucine-rich peptide named KLK & a synthetic oligonucleotide named ODN1a. The optimal molar ratio of KLK to ODN1a in mice is 25:1. AERAS-404 & saline placebo trial arms will be double-blinded since BCG causes a recognizable local injection site reaction, the BCG revaccination trial arm will be unblinded.
  Other Names: H4; H4:IC31
  Arms: AERAS-404 (15 mcgH4/500 nmol IC31)
Drug: Placebo — Saline
  Other Names: 0.9% Saline
  Arms: Placebo
Biological: Bacillus Calmette-Guérin (BCG) — BCG SSI Vaccine is registered in South Africa for prevention of TB in children and adults. BCG, an attenuated, live culture of the Bacillus Calmette-Guérin, was originally attenuated between 1906 and 1919 by serial passage of an M. bovis strain. The manufacturer Statens Serum Institut (SSI) in Copenhagen, Denmark derives this vaccine from the Danish BCG strain 1331. BCG SSI is supplied by the manufacturer in amber 10-dose vials containing 0.75 mg lyophilized SSI BCG. The BCG revaccination trial arm will be unblinded (open label).
  Other Names: BCG; BCG SSI
  Arms: Bacillus Calmette-Guérin (BCG)

SUMMARY:
Randomized, Placebo Controlled, Partially Blinded Phase II Study to Evaluate Safety, Immunogenicity, and Prevention of Infection with Mycobacterium tuberculosis of AERAS-404 and BCG Revaccination in Healthy Adolescents

DETAILED DESCRIPTION:
This Phase II, randomized, 3-arm, placebo controlled, partially blinded, clinical trial will be conducted in 990 healthy, HIV-uninfected, QFT-GIT negative, previously BCG vaccinated adolescents. The trial will be conducted at the South African Tuberculosis Vaccine Initiative (SATVI) site in the Western Cape region of South Africa, where epidemiological studies involving thousands of adolescents have been conducted over the last decade to characterize rates of Mtb infection and active TB disease in this age group. Subjects will be enrolled in two sequential cohorts and within each cohort subjects will be randomized in a 1:1:1 ratio to receive either AERAS-404 or saline placebo on Days 0 and 56, or BCG Vaccine SSI on Day 0. The first 90 subjects (30 from each arm) will form the Safety & Immunogenicity Cohort and will be subject to more intensive collection of safety data, with data reviewed by the Data Monitoring Committee (DMC), principal investigator and local medical monitor. Selected immunogenicity assays, including whole blood intracellular cytokine staining (ICS), will also be performed in this cohort. The remaining 900 subjects will be enrolled into the Correlates Cohort. All 990 subjects in the study will be evaluated for safety and biomarker outcomes, and for prevention of Mtb infection.

The primary Mtb infection endpoint will be QFT-GIT conversion from a negative to positive test, using the manufacturer's recommended threshold of 0.35 IU/mL, at any time-point after Day 84 and through end of follow-up for the primary endpoint. The 84-day 'wash-out' period is stipulated in order to exclude subjects who may have already been Mtb infected, but not yet converted their QFT-GIT test at screening, thus subjects who convert their QFT-GIT at Day 84 will not be included in the analyses of prevention of Mtb infection.

ELIGIBILITY:
Inclusion Criteria:

1. Has completed the written informed consent and assent process
2. Is age ≥ 12 years and ≤ 17 years on Study Day 0
3. Agrees to stay in contact with the study site for the duration of the study, provide updated contact information
4. For female subjects: agrees to avoid pregnancy from 28 days prior to Study Day 0 and for the full duration of the study.
5. Has general good health, confirmed by medical history and physical examination
6. Had BCG vaccination at least 5 years ago documented through medical history or by presence of healed BCG scar
7. Tests QFT-GIT negative at screening, using the manufacturer's recommended threshold of 0.35 IU/mL

Exclusion Criteria:

1. Acute illness on Study Day 0
2. Oral temperature ≥37.5°C on Study Day 0
3. Clinically significant (and no more than Grade 1 on the Toxicity Scale) abnormal laboratory values from blood collected within 21 days
4. Evidence of clinically significant (and no more than Grade 1 on the Toxicity Scale) systemic or local disease on urinalysis
5. History or evidence of any clinically significant systemic disease, or any acute or chronic illness that might affect the safety, immunogenicity, or efficacy of study vaccine in the opinion of the investigator
6. History of treatment for active TB disease or latent Mtb infection
7. History or evidence, including chest X-ray, of active TB disease
8. Shared residence with an individual receiving anti-TB treatment, or known incompletely treated culture or smear positive TB
9. History of autoimmune disease or immunosuppression
10. Used immunosuppressive medication within 42 days before Study Day 0
11. Received immunoglobulin or blood products within 42 days before Study Day 0
12. Received any investigational drug therapy or investigational vaccine within 182 days before Study Day 0
13. Received investigational TB vaccine, other than BCG
14. Planned administration/administration of a licensed vaccine in the period starting 28 days before and ending 28 days after each dose of study vaccine
15. History or laboratory evidence of any past or present possible immunodeficiency state not limited to any lab indication of HIV-1 infection
16. History of allergic disease likely to be exacerbated by any component of the study vaccine
17. History of alcohol or drug abuse
18. All female subjects: currently pregnant or lactating/nursing; or positive urine pregnancy test during screening
19. Received a (TST) within 3 months (90 days) prior to Study Day 0.
20. Any current medical, psychiatric, occupational, substance abuse problems problems that in opinion of investigator will make unlikely for the subject to comply with the protocol

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 989 (Actual)
Dates: Start 2014-02; Primary Completion 2017-08-28 (Actual); Study Completion 2017-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hatherill, MD, Principal Investigator — The South African Tuberculosis Vaccine Initiative(SATVI)
Locations (2):
- South Africa (2):
  - South African Tuberculosis Vaccine Initiative , Project Office, Brewelskloof Hospital , Harlem Street, Worcester, Cape Town, Western Cape
  - Desmond Tutu HIV Foundation (DTHF), Nyanga

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nemes E, Geldenhuys H, Rozot V, Rutkowski KT, Ratangee F, Bilek N, Mabwe S, Makhethe L, Erasmus M, Toefy A, Mulenga H, Hanekom WA, Self SG, Bekker LG, Ryall R, Gurunathan S, DiazGranados CA, Andersen P, Kromann I, Evans T, Ellis RD, Landry B, Hokey DA, Hopkins R, Ginsberg AM, Scriba TJ, Hatherill M; C-040-404 Study Team. Prevention of M. tuberculosis Infection with H4:IC31 Vaccine or BCG Revaccination. N Engl J Med. 2018 Jul 12;379(2):138-149. doi: 10.1056/NEJMoa1714021. PMID 29996082
- [Derived] Geldenhuys H, Mearns H, Miles DJ, Tameris M, Hokey D, Shi Z, Bennett S, Andersen P, Kromann I, Hoff ST, Hanekom WA, Mahomed H, Hatherill M, Scriba TJ; H4:IC31 Trial Study Group; van Rooyen M, Bruce McClain J, Ryall R, de Bruyn G; H4:IC31 Trial Study Groupa. The tuberculosis vaccine H4:IC31 is safe and induces a persistent polyfunctional CD4 T cell response in South African adults: A randomized controlled trial. Vaccine. 2015 Jul 9;33(30):3592-9. doi: 10.1016/j.vaccine.2015.05.036. Epub 2015 Jun 3. PMID 26048780

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AERAS-404 (15 mcgH4/500 Nmol IC31) | Bacillus Calmette-Guérin (BCG) | Placebo
Started | 330 | 330 | 329
Completed | 327 | 330 | 328
Not Completed | 3 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — participant refused to use contraception | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AERAS-404 (15 mcgH4/500 Nmol IC31) | Bacillus Calmette-Guérin (BCG) | Placebo | Total
Number analyzed (Participants) | 330 | 330 | 329 | 989
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 330 | 330 | 329 | 989
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (1.47) | 14.2 (1.49) | 14.3 (1.54) | 14.2 (1.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 162 | 169 | 520
  Male | 141 | 168 | 160 | 469
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 330 | 330 | 329 | 989
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 120 | 126 | 120 | 366
  White | 1 | 3 | 1 | 5
  More than one race | 208 | 200 | 207 | 615
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 330 | 330 | 329 | 989

OUTCOME MEASURES:

1. Primary Outcome: Safety Profile of H4:IC31 and BCG Revaccination in HIV-uninfected, Remotely BCG Vaccinated Adolescents.
Description: Number of unsolicited and solicited adverse events recorded post vaccination.
  Unsolicited adverse events: 28 days post each vaccination
  Solicited adverse events: 7 days post each vaccination (with diary cards used for 7 days after each vaccination for Safety and Immunogenicity Cohort only)
  Solicited and unsolicited injection site reaction adverse events: BCG Group - 84 days post vaccination; H4:IC31/Placebo Groups - 28 days post each vaccination
  Serious adverse events, adverse events of special interest, and SUSARs: Entire study period, with a minimum of 6 months following the last dose of study vaccine
Time Frame: Study day 7 thru 6 months after last vaccination
Measure: Number; unit: number of AEs
Arm/Group | AERAS-404 (15 mcgH4/500 Nmol IC31) | Bacillus Calmette-Guérin (BCG) | Placebo
Number analyzed (Participants) | 330 | 330 | 329
number of AEs | 286 | 1257 | 272

2. Primary Outcome: Number of Participants Testing Positive for Mtb at Day 84
Description: Rates of conversion to Mtb-positive measured by QuantiFERON-TB Gold In-tube (QFT-GIT) assay. The primary evaluation of Mtb infection was QFT-GIT conversion from a negative to positive test, using the manufacturer's recommended threshold of ≥0.35 IU/mL, at any time point after Day 84 and through end of follow-up for the primary endpoint. All participants with primary QFT-GIT conversion were followed for an additional 6 months post-conversion to ascertain the sustained QFT-GIT conversion and QFT-GIT reversion endpoints. Participants with an initial QFT-GIT conversion at Month 6 or 12 were asked to return for a final QFT-GIT evaluation and assessment for TB signs and symptoms at least 24 months after their initial vaccination.
  * H4:IC31 compared to placebo
  * BCG revaccination compared to placebo
Time Frame: Study day 84 through 6 months post-conversion
Population: Intent-to-Treat
Measure: Number; unit: participants
Arm/Group | AERAS-404 (15 mcgH4/500 Nmol IC31) | Bacillus Calmette-Guérin (BCG) | Placebo
Number analyzed (Participants) | 308 | 312 | 310
participants | 44 | 41 | 49

3. Secondary Outcome: Rates of Sustained Conversion to Mtb-positive
Description: Rates of sustained conversion to Mtb-positive as measured by QFT-GIT assay.
  * H4:IC31 compared to placebo
  * BCG revaccination compared to placebo
Time Frame: 6 months after initial conversion
Population: Modified Intent-to-Treat
Measure: Number; unit: participants
Arm/Group | AERAS-404 (15 mcgH4/500 Nmol IC31) | Bacillus Calmette-Guérin (BCG) | Placebo
Number analyzed (Participants) | 308 | 312 | 310
participants | 25 | 21 | 36

4. Secondary Outcome: Percentage of Participants With Immune Response to Vaccine in HIV-uninfected, Remotely BCG-vaccinated Adolescents: o H4:IC31 o BCG Revaccination
Description: A 13 color intracellular cytokine staining assay (ICS) was performed on peripheral blood mononuclear cells (PBMC) to assess CD4+ T cells that expressed IFN-γ, TNF, IL-2, IL-17, IL-22, CD107a, and/or CD154 alone or in combination in response to stimulation with peptide pools representing the entire amino acid sequence of the TB mycobacterial antigens Ag85B and TB10.4, and BCG antigens. Responders were IFN-gamma and/or IL-2 positive.
  An intracellular cytokine assay was performed on whole blood (WB) to measure the frequencies and patterns of CD4+ T cells expressing Th1 and Th17 cytokines following stimulation of whole blood with peptide pools representing the entire amino acid sequence of the TB mycobacterial antigens Ag85B and TB10.4, as well as viable BCG from the vaccine vial. Responders were IFN-gamma, IL-2, TNF, IL-17, and/or IL-22 positive.
Time Frame: Study day 70
Population: Modified ITT analysis set: Safety and immunogenicity cohort
Measure: Number; unit: percentage of participants
Arm/Group | AERAS-404 (15 mcgH4/500 Nmol IC31) | Bacillus Calmette-Guérin (BCG) | Placebo
Number analyzed (Participants) | 28 | 28 | 27
percentage of participants
  PBMC ICS: Percent of responders on day 70 | 81.8 | 16.0 | 12.0
  WB ICS: Percent responders on day 70 | 12.5 | 8.0 | 8.3

ADVERSE EVENTS:
Time Frame: Unsolicited AEs: 28 days post each vaccination Solicited AEs: 7 days post each vaccination (with diary cards used for 7 days after each vaccination for Safety and Immunogenicity Cohort only) Solicited and unsolicited injection site reaction AEs: BCG Group - 84 days post vaccination; H4:IC31/Placebo Groups - 28 days post vaccination Serious adverse events, adverse events of special interest, and SUSARs: Entire study period (minimum of 6 months following last dose of study vaccine)
Groups:
- Bacillus Calmette-Guerin (BCG): 1 Dose on Study Day 0
  Bacillus Calmette-Guérin (BCG): BCG SSI Vaccine is registered in South Africa for prevention of TB in children and adults. BCG, an attenuated, live culture of the Bacillus Calmette-Guérin, was originally attenuated between 1906 and 1919 by serial passage of an M. bovis strain. The manufacturer Statens Serum Institut (SSI) in Copenhagen, Denmark derives this vaccine from the Danish BCG strain 1331. BCG SSI is supplied by the manufacturer in amber 10-dose vials containing 0.75 mg lyophilized SSI BCG. The BCG revaccination trial arm will be unblinded (open label).
Arm/Group | AERAS-404 (15 mcgH4/500 Nmol IC31) | Bacillus Calmette-Guerin (BCG) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/330 | 0/330 | 1/329
Serious Adverse Events (participants affected / at risk) | 5/330 | 7/330 | 7/329
Other Adverse Events (participants affected / at risk) | 118/330 | 329/330 | 104/329
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AERAS-404 (15 mcgH4/500 Nmol IC31) (N=330) | Bacillus Calmette-Guerin (BCG) (N=330) | Placebo (N=329)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Near drowning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AERAS-404 (15 mcgH4/500 Nmol IC31) (N=330) | Bacillus Calmette-Guerin (BCG) (N=330) | Placebo (N=329)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 6 (7) | 5 (5)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 12 (15) | 10 (12) | 3 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 6 (6) | 3 (5) | 5 (7)
Fatigue (General disorders) | 16 (23) | 10 (15) | 18 (26)
Injection site erythema (General disorders) | 8 (9) | 0 (0) | 6 (7)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 34 (46) | 0 (0) | 20 (27)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 2 (2)
Injection site swelling (General disorders) | 15 (17) | 0 (0) | 8 (11)
Injection site warmth (General disorders) | 8 (12) | 0 (0) | 6 (10)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 2 (2) | 1 (1)
Vaccination site discharge (General disorders) | 0 (0) | 163 (169) | 0 (0)
Vaccination site discolouration (General disorders) | 0 (0) | 22 (22) | 0 (0)
Vaccination site erythema (General disorders) | 0 (0) | 147 (150) | 0 (0)
Vaccination site exfoliation (General disorders) | 0 (0) | 90 (92) | 0 (0)
Vaccination site induration (General disorders) | 0 (0) | 171 (171) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 45 (47) | 0 (0)
Vaccination site pallor (General disorders) | 0 (0) | 8 (8) | 0 (0)
Vaccination site papule (General disorders) | 0 (0) | 10 (10) | 0 (0)
Vaccination site pruritus (General disorders) | 0 (0) | 3 (3) | 0 (0)
Vaccination site scab (General disorders) | 0 (0) | 145 (147) | 0 (0)
Vaccination site scar (General disorders) | 0 (0) | 255 (255) | 0 (0)
Vaccination site swelling (General disorders) | 0 (0) | 172 (179) | 0 (0)
Vaccination site ulcer (General disorders) | 0 (0) | 104 (104) | 0 (0)
Vaccination site warmth (General disorders) | 0 (0) | 20 (22) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 2 (2)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 5 (5)
Rubella (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 31 (31) | 7 (7) | 26 (26)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Vaccination site pustule (Infections and infestations) | 0 (0) | 29 (29) | 0 (0)
Varicella (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 2 (2) | 4 (4)
Blood pressure increased (Investigations) | 2 (2) | 0 (0) | 3 (3)
Blood pressure systolic increased (Investigations) | 6 (6) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0) | 3 (3)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (2) | 3 (3)
Neutrophil count increased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Platelet count increased (Investigations) | 3 (3) | 2 (2) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 5 (5) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (5) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (22) | 7 (8) | 11 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1)
Headache (Nervous system disorders) | 25 (27) | 27 (32) | 31 (42)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (2) | 2 (2) | 4 (4)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3) | 2 (2) | 3 (4)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT02075203/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT02075203/SAP_001.pdf
  • Informed Consent Form (2014-01-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT02075203/ICF_002.pdf